CLINICAL TRIAL: NCT07178158
Title: Enhancing Addiction Treatment Through Psychoeducation: Evaluating the Feasibility and Acceptability of a Neuroscience-Informed Mobile App
Brief Title: Enhancing Addiction Treatment Through Psychoeducation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20032752
Record Dates: First submitted 2025-07-25; First posted 2025-09-17 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Substance Use Disorders
Keywords: tES/TMA: Transcranial electrical stimulation; CT: Cognitive Training; DASES: Drug Abstinence Self-Efficacy Scale
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: This is a pilot feasibility two-arm, randomized controlled study with parallel assignment and 1:1 allocation of individuals with SUDs who are currently in treatment to either (1) Intervention condition: NIPA + treatment as usual (TAU); or (2) Control condition: TAU only. The control condition (TAU) consists of medication treatment (buprenorphine) and group or individual behavior therapy. The intervention condition (NIPA+TAU) consists of TAU plus four ~20-minute long NIPA sessions, administered a week apart. Participants in both intervention and control conditions would undergo two phenotypic assessments on REDCap, one at baseline and one at the end of the intervention for the NIPA+TAU condition or at the end of week 4 for the TAU condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention condition (Experimental): The intervention condition consists of TAU plus four ~20-minute long NIPA sessions, administered a week apart (NIPA+TAU). Participants in both intervention and control conditions would undergo two survey assessments on REDCap, one at baseline and one at the end of the intervention for the NIPA+TAU condition or at the end of week 4 for the TAU condition.
  Interventions: Other: Installing the Metacognium software app
- Control condition (Placebo Comparator): The control condition consists of treatment as usual (TAU) consisting of medication treatment (buprenorphine) and group or individual behavior therapy. Participants in both intervention and control conditions would undergo two survey assessments on REDCap, one at baseline and one at the end of the intervention for the NIPA+TAU condition or at the end of week 4 for the TAU condition.
  Interventions: Other: Continue treatment as usual

INTERVENTIONS:
Other: Installing the Metacognium software app — Participants in the NIPA+TAU group will be sent two, URL's (one for iOS and one for Android) for installing the Metacognium software app, which hosts the four NIPA sessions. Participants will be provided with unique ID for registering and using the program on the Metacognium app. The NIPA sessions will be locked until participants have completed their baseline assessment. Once participants complete each NIPA session, they will receive an email and/or text notifying them that the next session is unlocked and that they can proceed to complete it.
  Arms: The intervention condition
Other: Continue treatment as usual — Continue your treatment schedule as usual with the for 4 weeks.
  Arms: Control condition

SUMMARY:
Addiction is a brain disorder characterized by a broad range of both apparent and subtle cognitive impairments in attention, memory, executive functions, and decision-making. These cognitive problems are clinically significant and may contribute to poor treatment outcomes in people with Substance Use Disorders (SUDs), such as a high risk of dropout, low treatment compliance, and shorter periods of abstinence. Studies on cognitive function in SUDs reveal that chronic use of drugs and alcohol can also negatively affect another crucial component of cognition: awareness, or metacognition. Metacognition is defined as an individual's ability to perceive and understand their cognitive functions and use this understanding to regulate them. One of the key consequences of metacognitive impairments is the lack of insight in people with SUDs, which adversely affects treatment outcomes. Substance users with poor metacognition are more reluctant to initiate or continue treatment and are more likely to deny their cognitive problems. Therefore, improving metacognition may remove or reduce motivational barriers to invest time and effort in the recovery process in general, and in the brain recovery process specifically. Despite the importance of neurocognition and metacognition in the recovery process for substance users, there is a dearth of interventions designed to target these functions.

DETAILED DESCRIPTION:
To address this gap, the Neuroscience-Informed Psychoeducation for Addiction (NIPA) program was developed as one of the first initiatives in the field of SUDs to raise individuals' awareness about cognitive deficits (metacognition) associated with drug and alcohol use. NIPA is an app-based digital program that integrates neuroscience-based psychoeducation and game-based cognitive training. It consists of four 20-minute-long sessions covering neurocognitive functions commonly impaired in SUDs, such as attention, memory, cognitive flexibility, and impulsivity / decision-making. Each session includes videos, animations and cartoons depicting specific cognitive problems (e.g. in attention, decision-making, etc.), followed by games created by adapting common neurocognitive tasks (e.g. Stroop task, gambling task), designed to engage the specific cognitive function reviewed in the session and to raise individual's awareness of how they employ these cognitive functions to solve game-based puzzles and real-life problems. Each cognitive function is depicted in terms of the underlying brain network(s) (e.g. default mode network, salience network), which is followed by a set of brain training strategies and exercises that aim to improve resilience when exposed to substances and to motivate patients to invest time and effort in their treatment and to pursue cognitive rehabilitation interventions. The main goals of the proposed study are to determine whether the intervention is feasible and acceptable for patients with SUDs who are currently in treatment; and to obtain some preliminary data on its utility to increase metacognitive awareness, reduce depression and anxiety, and improve daily executive functioning and impulse control in patients with SUDs. We hypothesize that providing patients with the NIPA program may improve their metacognition, daily executive function, and mental health.

ELIGIBILITY:
Inclusion Criteria:

* current DSM-5 opioid and/or stimulant use disorder
* currently on medication treatment for SUD
* owning a smartphone with sufficient functionality to download and utilize the NIPA app.

Exclusion Criteria:

* current psychosis, mania, or suicidal/homicidal ideation
* non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruiting for the Neuroscience-Informed Psychoeducation for Addiction (NIPA) intervention | Baseline through 4 week intervention
  The recruitment rate is quantified as the % of all participants who satisfy the inclusion criteria and agree to participate.
Retention/adherence rate for the Neuroscience-Informed Psychoeducation for Addiction (NIPA) Intervention | Baseline through 4 week intervention
  Retention/adherence rate is quantified as the % of participants who remain enrolled until the end of the study, completing all NIPA sessions and pre- and post-assessments.
Completion rate for the Neuroscience-Informed Psychoeducation for Addiction (NIPA) intervention | Baseline through 4 week intervention
  Completion rate, indexing the number of training sessions completed by each participant.
Measure acceptability of the Neuroscience-Informed Psychoeducation for Addiction (NIPA) intervention | Baseline through 4 week intervention
  Acceptability is measured with a 10-item questionnaire that uses a 10-point Likert scale, with higher scores indicating greater acceptability. Items include perceived enjoyment, convenience, informativeness, applicability, effectiveness, satisfaction, continued use, barriers to use, and most/least liked aspects.

SECONDARY OUTCOMES:
Assess Drug Knowledge | Baseline through 4 week intervention
  Drug knowledge is assessed using a questionnaire developed by our team. The questionnaire consists of 12 true-or-false items adapted from the psychoeducational materials provided in the program. Participants will complete the questionnaire at baseline before the intervention, and again after the intervention ends. Drug knowledge scores will be calculated as the total number of true responses and reported as both numbers and percentages.
Measure attitudes towards drugs and alcohol | Baseline through 4 week intervention
  The Attitudes Toward Alcohol Use Scale and the Attitudes Toward Drug Use Scale each consist of four items. Intentions for use will be measured by asking participants to rate their intention to use various substances in the next six months on a 7-point Likert scale. Higher scores indicate greater intention to use. The scales evaluate participants' consideration of being under the influence of the respective substances. Participants complete the questionnaire at baseline, prior to the intervention, and again after the intervention has concluded. Attitudes toward drugs and alcohol will be reported using the mean and standard deviation.
Intention for Substance Use | Baseline through 4 week intervention
  Intention to use drugs and alcohol will be measured by asking participants to rate their intention to use various substances in the next month on a 7-point Likert scale, Higher scores indicate greater intention to use. Participants will complete the questionnaire at baseline prior to the intervention, and again after the intervention ends. Intentions to use will be reported using the mean and standard deviation.
Metacognitive Awareness | Baseline through 4 week intervention
  The 15-item Mindful Attention Awareness Scale will measure metacognitive awareness. Each item is rated on a 6-point Likert scale, with higher total scores reflecting greater levels of mindfulness and awareness. Participants will complete the questionnaire at baseline before the intervention, and again after the intervention ends. The metacognitive awareness total score will be reported using the mean and standard deviation.

OTHER OUTCOMES:
Negative Affect-Anxiety | Baseline through 4 week intervention
  Anxiety will be measured using the PROMIS Anxiety Scale, a 4-item measure of emotional distress related to fear, anxious misery, hyperarousal, and associated somatic symptoms experienced over the past 7 days. Each item is rated on a 5-point Likert scale, reflecting the frequency of the symptoms. Higher scores indicate more severe symptoms. Participants will complete the questionnaire at baseline, before the intervention, and again after the intervention ends. Anxiety total score will be reported using the mean and standard deviation.
Negative Affect- Depression | Baseline through 4 week intervention
  Depression will be measured using the PROMIS Depression Scale, a 4-item measure of negative mood, self-perception, social cognition, and reduced positive affect and engagement. It measures the frequency of each symptom using a 5-point Likert scale. Higher scores indicate more severe symptoms. Participants will complete the questionnaire at baseline, before the intervention, and again after the intervention ends. Depression total score will be reported using the mean and standard deviation.
Drug Abstinence Self-efficacy | Baseline through 4 week intervention
  The Drug Abstinence Self-Efficacy Scale is a 20-item scale that will be used to measure a participants confidence to remain abstinent from alcohol and drug use in situations that elicit drinking or substance use cues. It consists of four subscales measuring types of relapse precipitants such as negative affect, positive social, physical, and other concerns, and withdrawal and urges, measured on a 5-point Likert scale, with higher scores indicating greater self-efficacy to resist substance use in challenging situations. Participants will complete the questionnaire at baseline prior to the intervention, and again after the intervention ends. Self-efficacy total score will be reported using the mean and standard deviation.
Barkley Deficits in executive functioning | Baseline through 4 week intervention
  The Barkley Deficits in Executive Function Scale will be used to measure subjective deficits in executive functioning as they manifest in daily life, using a 4-point Likert scale. Higher scores indicate greater executive function deficits. Participants will complete the questionnaire at baseline, prior to the intervention, and again after the intervention ends. Deficits in executive functioning total score will be reported using the mean and standard deviation
Delay Discounting | Baseline through 4 week intervention
  The Monetary-Choice Questionnaire, consisting of 27 items, will be used to assess delay discounting. The participant chooses between a smaller, immediate (hypothetical) monetary reward and a larger, delayed monetary reward. These choices are used to calculate a discounting rate parameter (k). Higher k values indicate a stronger preference for immediate rewards and thus greater impulsivity. Participants will complete the questionnaire at baseline before the intervention, and again after the intervention ends. Discounting rate (K) score will be reported using the mean and standard deviation. Parametric t-test or nonparametric Mann-Whitney U test to examine between-group differences, and paired t-test or non-parametric Wilcoxon signed-rank test to determine if the within-individual change in the group is statistically significant. Pre-existing differences in all measures collected at baseline will be controlled in subsequent analyses, using baseline scores as covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Jasmin Vassileva, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rezapour T, McLean KL, Psederska E, Maleki KN, Ekhtiari H, Vassileva J. Neuroscience-informed psychoeducation for addiction: a conceptual and feasibility study. Front Psychiatry. 2025 Feb 12;16:1527828. doi: 10.3389/fpsyt.2025.1527828. eCollection 2025. PMID 40012711
- [Background] Barkley, RA. Barkley Deficits in Executive Functioning Scale (BDEFS) New York, NY: The Guilford Press; 2011.
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Heckman CJ, Dykstra JL, Collins BN. Substance-Related Knowledge, Attitude, and Behavior among College Students: Opportunities for Health Education. Health Educ J. 2011 Dec;70(4):383-399. doi: 10.1177/0017896910379694. PMID 22303033
- [Background] Hiller ML, Broome KM, Knight K, Simpson DD. Measuring self-efficacy among drug-involved probationers. Psychol Rep. 2000 Apr;86(2):529-38. doi: 10.2466/pr0.2000.86.2.529. PMID 10840908
- [Background] Khazaee-Pool M, Naghibi SA, Pashaei T, Chaleshgar-Kordasiabi M, Daneshnia M, Ponnet K. Drug Abstinence Self-Efficacy Scale (DASES): psychometric properties of the Farsi version. Subst Abuse Treat Prev Policy. 2021 Jan 3;16(1):1. doi: 10.1186/s13011-020-00336-9. PMID 33388062
- [Background] Kirby, K. N., Petry, N. M., & Bickel, W. K. (2012). Monetary Choice Questionnaire [Dataset]. https://doi.org/10.1037/t10044-000
- [Background] Lins de Holanda Coelho G, H P Hanel P, Vilar R, P Monteiro R, Gouveia VV, R Maio G. Need for Affect and Attitudes Toward Drugs: The Mediating Role of Values. Subst Use Misuse. 2018 Nov 10;53(13):2232-2239. doi: 10.1080/10826084.2018.1467454. Epub 2018 May 4. PMID 29727251
- [Background] Manser P, Poikonen H, de Bruin ED. Feasibility, usability, and acceptance of "Brain-IT"-A newly developed exergame-based training concept for the secondary prevention of mild neurocognitive disorder: a pilot randomized controlled trial. Front Aging Neurosci. 2023 Sep 21;15:1163388. doi: 10.3389/fnagi.2023.1163388. eCollection 2023. PMID 37810620
- [Background] Meredith LR, Maralit AM, Thomas SE, Rivers SL, Salazar CA, Anton RF, Tomko RL, Squeglia LM. Piloting of the Just Say Know prevention program: a psychoeducational approach to translating the neuroscience of addiction to youth. Am J Drug Alcohol Abuse. 2021 Jan 2;47(1):16-25. doi: 10.1080/00952990.2020.1770777. Epub 2020 Jul 20. PMID 32687415
- [Background] Schalet BD, Pilkonis PA, Yu L, Dodds N, Johnston KL, Yount S, Riley W, Cella D. Clinical validity of PROMIS Depression, Anxiety, and Anger across diverse clinical samples. J Clin Epidemiol. 2016 May;73:119-27. doi: 10.1016/j.jclinepi.2015.08.036. Epub 2016 Feb 27. PMID 26931289
- See also: Article full text — https://doi.org/10.3389/fpsyt.2025.1527828